CLINICAL TRIAL: NCT06902233
Title: High-definition Transcranial Infraslow Gray Noise Stimulation for Treatment of Chronic Low Back Pain: A Double-blinded Randomised Controlled Clinical Trial.
Brief Title: Brain Network Stimulation for Chronic Low Back Pain.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Otago (Other)
Collaborators: Dunedin School of Medicine, University of Otago, Dunedin, New Zealand (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024 FULL 21891; 24-176 (Other Grant/Funding Number: Health Research Council of New Zealand)
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: Chronic low back pain; Brain stimulation; Transcranial infraslow grey noise stimulation; Randomised controlled trial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The statistician analysing the data will also be blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High definition transcranial infraslow gray noise stimulation (HD-tIGNS) (Experimental): For the active stimulation group, the HD-tIGNS will be delivered for 30min, with 60s ramp up and ramp down at the beginning and end of each stimulation session, with continuous stimulation in between. The gray noise (50%) will be superimposed on the infraslow (0.1Hz) sinusoidal waveform (50%), with the maximum current strength of 2.0 mA per electrode and the maximum total current injected being 4.0mA.
  Interventions: Device: High-definition transcranial infraslow grey noise stimulation
- Sham stimulation (Sham Comparator): For the sham stimulation group, to create an identical skin sensation to the active stimulation, we will use the Actisham protocol (with FC2 as the itchy electrode) created by the Neuroelectrics. The current will be applied for a 5s ramp up and 5s ramp down at the beginning of each stimulation session, without any current for the remainder of the stimulation period. The sham session will last as long as the HD-tIGNS session to blind the procedure appropriately.
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: High-definition transcranial infraslow grey noise stimulation — HD-tIGNS will be administered three times a week (30 minutes/ session) for a total of 4 weeks (i.e., 12 sessions in total) using a 32-channel transcranial current stimulator. The HD-tIGNS will be used to alter the functional connectivity strength between the three cortical networks [namely the salience network (SN), the default mode network (DMN) and the somatomotor network (SMN)] in the infraslow frequency spectrum (0.1 Hz). A total of fifteen circular Ag/AgCl electrodes [eleven stimulation electrodes (C1, C2, C3, C4, F7, F8, FC3, FT7, FPz, Fz, and O2) and four electrodes with zero current (FC1, FC2, FC4, and FCz)] will be placed on a neoprene head cap following the International 10-10 EEG system. The optimal montages has been created using the Stimweaver optimization software by the Neuroelectrics company, to specifically decrease the functional connectivity i.e., phase synchronization of the brain regions of the SN with the SMN and the DMN.
  Arms: High definition transcranial infraslow gray noise stimulation (HD-tIGNS)
Device: Sham Comparator — The Actisham protocol (with FC2 as the itchy electrode) created by the Neuroelectrics will be used for the sham stimulation group. Similar to the active treatment group, the actisham will be administered three times a week (30 minutes/ session) for a total of 4 weeks (i.e., 12 sessions in total) using a 32-channel transcranial current stimulator.Similar to active group, a total of fifteen circular Ag/AgCl electrodes will be placed on a neoprene head cap following the International 10-10 EEG system to appropriately blind the participant. The electrodes would comprise of four stimulation electrodes (FC1, FC2, FC4, and FCz) and eleven electrodes (C1, C2, C3, C4, F7, F8, FC3, FT7, FPz, Fz, and O2) with zero current.
  Other Names: Sham stimulation; Actisham stimulation
  Arms: Sham stimulation

SUMMARY:
This study looks at the non-invasive brain stimulation technique in people with chronic low back pain to see:

* How effective non-invasive brain stimulation is at improving pain intensity in people with chronic low back pain?
* How safe non-invasive brain stimulation is and what side effects there may be?
* What study participants think of the study procedures and of the non-invasive brain stimulation as a treatment technique for chronic low back pain.

Participants will be assigned to receive either active brain stimulation group or sham stimulation group randomly.

Participants will be required to attend a total of twelve treatment sessions (approximately 1-hour each, three sessions per week, for four consecutive weeks).

Assessments will be done at baseline (in the week 0), immediately post-completion of the intervention (in the week 5), and at the follow-up of one-month (in the week 8), three-months (in the week 16) and six-months (in the week 28) post-completion of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 75 years on the day of screening
* Pain in the lower back (region between 12th rib and gluteal fold) with or without accompanying leg pain that occurs for at least half the days in the last six months
* An average pain intensity of ≥4 on the 11-point NPRS (0=No pain to 10=Pain as bad as you can imagine) in the week prior to enrolment
* A disability score of ≥5 on Roland-Morris Disability Questionnaire (RMDQ).

Exclusion Criteria:

* Known or suspected serious spinal pathology (fracture; lumbar canal stenosis, malignant, inflammatory or infective diseases of the spine; cauda equina syndrome or widespread neurological disorder)
* Suspected or confirmed pregnancy or less than six months post-partum
* Inflammatory disorders
* Auto-immune conditions
* Recent soft tissue injuries of the back in the last 3 months
* Recent steroid injections to the back in the past 3 months
* Recent spinal surgery in the past 12 months or scheduled/waiting for any major surgical procedures during the treatment or follow-up period or underwent rhizotomy or any neurosurgical procedures
* History of neurological conditions, or psychiatric disorders (except depression and anxiety disorders)
* History of cancer, or currently receiving/scheduled for receiving therapy for cancer
* Cognitive impairments (dementia, Alzheimer's disease; indicated by a total score of 24 or below on Mini-Mental State Examination)
* Alcohol or substance abuse
* History of epilepsy or seizures
* Presence of any electronic implants (e.g., pacemaker), metal implant in the body (particularly head and neck), or spinal cord stimulator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | The primary endpoint for efficacy assessment of HD-tIGNS will be change in the average pain intensity over the past week from baseline to one-week post completion of treatment.
  Average pain intensity over the past week measured on a numeric pain rating scale (NPRS) of 0 to 10 (0=No pain to 10=Pain as bad as you can imagine) from the Brief Pain Inventory short form

SECONDARY OUTCOMES:
Pain intensity | Change in the average pain intensity over the past week from baseline to one-month, three-months and six-months post completion of treatment.
  Average pain intensity over the past week measured on a NPRS of 0 to 10 (0=No pain to 10=Pain as bad as you can imagine) from the Brief Pain Inventory short form.
Pain interference | Change in the pain interference from baseline to one-week, one-month, three-months and six-months post completion of treatment.
  Brief Pain Inventory (BPI), a standardised, validated questionnaire, will be used to capture pain interference in daily activities
Pain unpleasantness | Change in the pain unpleasantness from baseline to one-week, one-month, three-months and six-months post completion of treatment.
  Pain unpleasantness (affective component) in past one week measured on an 11-point NPRS-unpleasantness scale.
Pain Bothersomeness | Change in the pain bothersomeness from baseline to one-week, one-month, three-months and six-months post completion of treatment.
  Pain bothersomeness in past one week measured on an 11-point NPRS-bothersomeness scale.
Patient global impression of change | Recorded at one-week, one-month, three-months, and six-months post completion of treatment.
  Patient global impression of change (PGIC) 7-point scale will be used to evaluate participants perception of overall improvement compared to baseline.
Movement Evoked Pain: Repeated spinal bending | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment.
  Participants will be asked to perform 20 repetitions each of 2 repeated spinal bending tasks (forward and backward bending) independently, with at least a 10-15 minute rest in between. Participants will rate their pain intensity on a NPRS (0=no pain to 100=worst pain imaginable) before commencing the movements, then following every 5 repetitions.
Movement Evoked Pain: Back Performance scale | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment.
  Back Performance scale (BPS) will be used to assess movement evoked pain (MEP) intensity during five functional tasks. Participants will be asked to rate their "pain rating at worst" during each task on a 0 to 100 NPRS. An MEP intensity composite score will be calculated by averaging pain ratings for the 5 tasks, with higher scores indicating greater MEP intensity.
Mechanical temporal summation | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment.
  Mechanical temporal summation (MTS): will be assessed using a nylon monofilament (Semmes monofilament 6.65, 300 g) at the most painful low back region (nominated by the participant) and the non-dominant wrist (distant region). Brief 10 repetitive contacts will be delivered at a rate of 1 Hz, externally cued by auditory stimuli. Participants will be asked to rate the level of pain experienced on NRS (0=no pain to 100=extreme pain) immediately after the first contact and to rate their greatest pain intensity after the 10th contact; with the difference representing the maximum amount of MTS across 10 contact points. Average of three trials will be calculated, with a positive score indicating an increase in MTS. The MTS index will be defined as the ratio of 'follow-up' pain rating divided by 'baseline' pain rating.
Pressure Pain Threshold | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment.
  Pressure pain threshold (PPT) will be assessed over the most painful low back region (nominated by the participant) and the non-dominant wrist (distant region) using a computerized, handheld digital algometer (AlgoMed; Medoc, Ramat Yishai, Israel) probe pressed over marked test site at a rate of 30 kPa/s. Participants will press the algometer trigger button in the patient control unit when pressure sensation changes to first pain. Average of three trials will be calculated and used for analysis
Function | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment.
  Roland-Morris Disability Questionnaire (RMDQ) will be used to assess self-reported functional abilities; within-group MCID is 30% decrease from baseline.
Health Related Quality of Life | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment.
  European Quality of Life-5 Dimensions scale will be used to assess the health-related quality of life; within-group MCID is 0.03 and 10.5 from baseline for the health index and the thermometer respectively.
Well-Being | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment.
  World Health Organization- Five Well-Being Index (WHO-5) will be used to measure the participant's current mental wellbeing.
Depression | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment.
  Depression and Somatic Symptoms Scale (DSSS) will be used to evaluate the severity of depression (cutoff score of ≥15).
Catastrophizing | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment.
  Pain Catastrophizing Scale (PCS) will be used to measure the extent of catastrophic thoughts and feelings about their pain.
Attention to pain | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment.
  Pain Vigilance and Awareness Questionnaire (PVAQ) will be used to measure the frequency of habitual 'attention to pain' over the past two weeks.
Positive and Negative Affect | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment.
  Positive and Negative Affect Schedule (PANAS-short form) will be used to measure the two-dominant dimensions of affect style, positive and negative affect.
Self-efficacy | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment.
  Pain self-efficacy (PSE), a 2-item questionnaire, will be used to assess pain self-efficacy beliefs.
Intolerance to Uncertainity scale short form | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment.
  Intolerance of uncertainty (IUS) scale- short form (12 item), will be used to assess how individuals perceive and respond to uncertainty in their daily lives. Total score ranges between 5 to 60 with higher scores indicating higher levels of intolerance to uncertainity.
Tampa scale of Kinesiophobia | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment.
  Tampa Scale of Kinesiophobia (TSK-11), will be used to quantify fear of movement. The scores ranges from 11 to 44, where higher scores indicate greater fear of pain, movement, and injury.
Rescue analgesics / Concomitant treatment | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment. QAQ will also be collected during intervention period, either at start of sessions (S1, S4, S7, S10) or after completion of the session (S12).
  The Quantitative analgesic questionnaire (QAQ) will be used to capture daily medication usage and a score will be generated to calculate weekly average pain medication use throughout the study. Other concomitant treatments including exercises, healthcare visits, etc. with the type and dosage will also be recorded throughout the study period using a diary.
Electroencephalography | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment. EEG will also be collected during intervention phase either at start of the sessions (S1,S4,S7,S10) or after completion of sessions (S1 and S12).
  Resting-state eyes closed electroencephalogram (EEG) (~10 minutes) will be obtained using SynAmps RT Amplifier (Compudemics Neuroscan) with 64 electrodes placed in the standard 10-10 International placement. During the intervention phase, resting state EEG will be collected using the Neuroelectrics Starstim32 system.
  Exact low-resolution brain electromagnetic tomography (eLORETA), will be used through the LORETA-key software package to estimate the intracerebral electrical sources that generate scalp-recorded electrical activity. Lagged phase synchronization will be used as a measure of functional connectivity and will be calculated between the targeted brain regions (i.e., dorsal anterior cingulate cortex, Somatosemsory cortex, motor cortex, Insula, pregenual anterior cingulate cortex) in the infraslow frequency band (0.1Hz).
Emotional Stroop Task | Recorded at baseline, and at one-week, one-month, three-months, and six-months post completion of treatment. Stroop testing will be also be done during the intervention phase either at start of sessions (S4, S7, S10) or after completion of session (S12).
  Participants will be presented with words from 3 interference categories (Sensory pain-related, Affective pain-related, and Positive-emotional) and 3 control categories (comprising of matched neutral words) in four different colours (blue, red, yellow, green) and will be asked to press one of four response keys to indicate the colour of the words regardless of their meaning. The participant's response, the correctness of the response, and the response latency (in ms) of each of the 6 different categories will be recorded. Each word will be displayed for 1.5s and there will be 16 words in a 24s block. A single trial will be conducted, and it will include 16 blocks, i.e., 2 blocks for each word-type, 2 blocks for each corresponding control word set, and four fixation-cross (rest) blocks (24s duration) presented on the screen at the beginning and twice within a trial. The average of two test blocks will be calculated and used for analysis.

OTHER OUTCOMES:
Safety of the intervention | Recorded at all the intervention sessions and at one-week, one-month, three-months and six-months post-completion of intervention.
  Discontinuation-Emergent Sign and Symptom checklist will be used to record worsening or improvement of the side effects compared with status prior to previous session.

CONTACTS AND LOCATIONS:
Overall Officials: Divya Adhia, Ph.D, Principal Investigator — Department of Surgical Sciences, Dunedin School Of Medicine, University of Otago, Dunedin, New Zealand.
Locations (1):
- Department of Surgical Sciences, Dunedin School of Medicine, University of Otago, Dunedin, Otago, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
All anonymised participant data will be available from the Principal Investigator upon reasonable request for future research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD will be available after completion of the data collection phase i.e., approximately from January 2028, until 10 years after completion of the study (approximately January 2038).
Access Criteria: All supporting information will be published in a peer-reviewed journal.
  The anonymous IPD will be available from the Principal Investigator upon reasonable request for future research.

REFERENCES:
- [Derived] Adhia DB, Mani R, Reynolds J, Glue P, Potiki J, Vanneste S, De Ridder D. Functional connectivity-targeted high-definition transcranial infraslow grey noise stimulation for chronic low back pain: protocol for a double-blinded, randomised, controlled clinical trial. BMJ Open. 2025 Aug 24;15(8):e103019. doi: 10.1136/bmjopen-2025-103019. PMID 40850927

DOCUMENTS (1):
  • Informed Consent Form (2024-11-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT06902233/ICF_000.pdf